CLINICAL TRIAL: NCT03522818
Title: Enuresis Alarm - Is a Manual Trigger System Beneficial?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gina Lockwood (Other)
Collaborators: PottyMD (Unknown)
Responsible Party: Sponsor-Investigator, Gina Lockwood, Principal Investigator, Medical Doctor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201801703
Record Dates: First submitted 2018-03-16; First posted 2018-05-11 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Enuresis, Nocturnal
MeSH Terms: conditions — Nocturnal Enuresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal (Active Comparator): Group will use the alarm as provided by the manufacture.
  Interventions: Behavioral: Normal
- Manual trigger (Experimental): Group will use the same model but will be instructed to manually trigger the alarm 1-2 hours after the child falls asleep.
  Interventions: Behavioral: Manual Trigger

INTERVENTIONS:
Behavioral: Manual Trigger — Will use the alarm as provided by the manufacture but parent has to manual trigger the alarm 1-2 hours after the child falls asleep.
  Arms: Manual trigger
Behavioral: Normal — Will use the alarm as provided by the manufacture.
  Arms: Normal

SUMMARY:
The purpose of this study is to evaluate whether the bedwetting alarm trigger activated by parents to wake their child, in addition to the moisture alarm, will improve treatment success compared to the moisture alarm alone.

DETAILED DESCRIPTION:
Nocturnal enuresis is a common issue in children, and use of bedwetting alarms has shown the best long-term success. However, use of alarms is very time-intensive, often taking months before yielding results. Researchers in the division of pediatric urology are initiating a randomized controlled study comparing a standard bedwetting alarm with a newly developed technology, with the hope that the new alarm will result in better, more rapid, and easier treatment for bedwetting.

Children between the ages of 5 to 15 years old who have issues with bedwetting after successful toilet training may qualify for the study.

Participants must first be evaluated by a pediatric urology specialist.

ELIGIBILITY:
Inclusion Criteria:

* children ages 5-15 years
* Diagnosis of Primary Monosymptomatic Nocturnal Enuresis
* >2 wet nights per week
* Score of 7 or below on questions 1-6 and 9-13 on Vancouver Dysfunctional Elimination Questionnaire
* Patients/parents compliance in recording data > 50% of nights

Exclusion Criteria:

* Known comorbid conditions: daytime incontinence, anatomic abnormalities (hydronephrosis, VUR), recurrent urinary tract infection, dysuria, neurogenic bladder, developmental delay, encopresis, diabetes insipidus, previous history of urologic surgery
* Concomitant DDAVP use, anticholinergic use, B3 agonist use

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2018-03-09 (Actual); Primary Completion 2023-03-12 (Estimated); Study Completion 2023-09-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the change and % reduction in mean number wet nights/week (>90%, 50-89%, <50%) of patients with treatment success with use of a manual trigger + moisture alarm vs. moisture alarm only | one year
  Bladder Diary (Participant self-reported)

CONTACTS AND LOCATIONS:
Overall Officials: Gina M Lockwood, MD, MS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No